CLINICAL TRIAL: NCT04851379
Title: PLACE OF THE 18F-FDG-PET/CT IN THE DIAGNOSTIC WORKUP IN PATIENTS WITH CLASSICAL FEVER OF UNKNOWN ORIGIN (FUO)
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0187
Record Dates: First submitted 2021-04-13; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Fever of Unknown Origin
Keywords: Fever of Unknown Origin; 18F-FDG-PET/CT
MeSH Terms: conditions — Fever of Unknown Origin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective : To explore the diagnostic contribution of the 18F-FDG-PET/CT in a population of patients with classical fever of unknown origin (FUO), to precise its place in the diagnostic decision tree in a real-life setting and to identify factors associated with a diagnostic 18F-FDG-PET/CT.

Methods: All adult patients (age≥18 years) with a diagnosis of classical FUO who underwent a 18F-FDG-PET/CT in the University Hospital of Montpellier (France) between April 2012 and December 2017 were included. True positive 18F-FDG-PET/CT which evidenced a specific disease causing FUO were considered to be contributive.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* a diagnosis of classical FUO who underwent a 18F-FDG-PET/CT

Exclusion Criteria:

-refusal to participate-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study included all adult patients (age≥18 years) with a diagnosis of classical FUO who underwent a 18F-FDG-PET/CT in the University Hospital of Montpellier (France) between April 2012 and December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
the diagnostic contribution of the 18F-FDG-PET/CT | day 1
  the diagnostic contribution of the 18F-FDG-PET/CT in a population of patients with classical FUO.

SECONDARY OUTCOMES:
18F-FDG-PET/CT place in the diagnostic decision tree in a real-life setting | day 1
  18F-FDG-PET/CT place in the diagnostic decision tree in a real-life setting
factors associated with a diagnostic 18F-FDG-PET/CT. | day 1
  factors associated with a diagnostic 18F-FDG-PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Camille ROUBILLE, MCUPH, Study Director — UH MONTPELLIER
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
nc